CLINICAL TRIAL: NCT04431089
Title: A Phase II Multicenter Study to Investigate the Efficacy and Safety of SHC014748M in Patients With Relapsed or Refractory Follicular (FL) or Marginal Zone (MZL) Lymphoma
Brief Title: Efficacy and Safety of SHC014748M in Patients With Relapsed or Refractory Follicular (FL) or Marginal Zone (MZL) Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHC014-II-01
Record Dates: First submitted 2020-06-01; First posted 2020-06-16 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-06

CONDITIONS: Follicular Lymphoma(FL); Marginal Zone Lymphoma(MZL)
Keywords: FL; MZL; SHC014748M; Phosphatidylinositol 3-kinase (PI3K)
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHC014748M treatment (Experimental): SHC014748M capsule, 200mg QD, 28 days for each cycle
  Interventions: Drug: SHC014748M

INTERVENTIONS:
Drug: SHC014748M — Each treatment cycle is comprised of 28-day consecutive dosing of SHC014748M, 200mg QD (Days 1 to28). Upon completion of each cycle, patients may continue to receive oral SHC014748M if they can benefit from the treatment and the toxicity is tolerable.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SHC014748M in patients with relapsed or refractory relapsed or refractory follicular (FL) or marginal one (MZL) lymphoma.

DETAILED DESCRIPTION:
This is a phase II, multicenter study to assess the efficacy and safety of SHC014748M, an oral inhibitor of PI3K delta, in patients with relapsed or refractory relapsed or refractory follicular (FL) or marginal one (MZL) lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Adult, male and female volunteers, above 18 years of age inclusive.
* Histologically or cytologically confirmed diagnosis of relapsed or refractory FL(grade 1, 2 or 3a) and MZL, including splenic marginal zone lymphoma(SMZL), nodal marginal zone B cell lymphoma(NMZL) and mucosa associated lymphoid tissue(MALT) lymphoma. Relapse refers to disease progression after adequate treatment to remission；refractory refers to no remission after adequate treatment. The above "remission" includes complete remission and partial remission. Adequate treatment refers to two or more treatments with CD20 monoclonal antibody (CDE approved for marketing) combined with alkylation agent, including but not limited to bendamustine, cyclophosphamide, ifosfamide, chlorambucil, melphalan, busulfan and nitrosoureas.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
* Life expectancy ≥ 3 months.
* Patients have at least 1 measurable lesion that measures ≥1.5 cm in a single dimension as assessed by CT or MRI.
* Adequate organ function, as defined by the following values:ANC≥1.0×10^9/L； PLT≥50×10^9/L;Hb≥80 g/L;TBIL≤2×ULN(TBIL>2×ULN for subjects with Gilbert syndrome,TBIL>3×ULN for subjects with focal compression of bile duct judged by investigators); ALT and AST≤2.5×ULN(ALT and AST≤5×ULN for subjects with impaired liver function caused by hepatic infiltration);blood urea nitrogen(BUN) and Cr≤1.5×ULN;LVEF≥50%;QTcF <450 ms for male, QTcF <470 ms for female.
* Men and women of childbearing potential are willing to employ an effective method of contraception for the entire duration of study and 6 months after the last dose, and female subjects of childbearing potential have a negative pregnancy test at baseline.
* Subjects did not participate in other clinical trials within 1 month prior to study entry.
* Provision of signed and dated, written informed consent prior to any study-specific evaluation.

Exclusion Criteria:

* Previous treatment with any PI3Kδ inhibitors.
* Evidence of aggressive lymphoma(suspected clinical transformation should be conformed by biopsy).
* Had any other anti-tumor treatment within 4 weeks prior to screening(including radiotherapy, chemotherapy, Chinese herbal anti-tumor treatment and major surgery); targeted therapy with 5 half-life period prior to screening.
* Evidence of central nervous system involvement of the malignancy.
* Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, uncontrolled pleural effusion and ascites, uncontrolled diabetes, severe or debilitating lung disease.
* Any of the severe heart diseases, including New York Heart Association (NYHA) Class II or greater heart failure, arrhythmias requiring medical treatment, and history of myocardial infarction or unstable angina within 6 months prior to screening.Requiring any concomitant medication known to prolong the QT interval within 5 half-life period.
* Evidence of active bacterial, fungal, or viral infection, and need systemic treatment.
* Active infection with hepatitis B virus (HBV) (HBsAg positive, or HBsAg negative and HBV-DNA positive), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* Concomitant use of any strong inhibitors or inducers of CYP3A4(except drug withdrawal prior to first dose of investigational drug.
* Use of granulocyte colony-stimulating factor(G-CSF) or blood transfusion within 7 days before the hematology test at screening.
* Prior autologous hematopoietic stem cell transplantation within 3 months prior to screening.
* History of immune deficiency(acquired and congenital), or history of organ transplantation, or allogeneic bone marrow or hematopoietic stem cell transplantation; with active autoimmune disease or history of autoimmune disease including Interstitial pneumonia, autoimmune enteritis, autoimmune hepatitis and systemic lupus erythematosus
* History of any uncured malignant tumor in the past five years except for the following: clinically cured cervical or breast carcinoma in situ, local basal cell or squamous cell carcinoma of the skin, thyroid tumor.
* Inability to swallow the drug, or history of diseases affecting gastrointestinal functions significantly including malabsorption syndrome,bariatric surgery,inflammatory bowel disease, partial or complete intestinal obstruction.
* Adverse events occurred during previous anticancer therapy have not been recovered to ≤1(CTCAE 5.0).
* History of hypersensitivity to the main composition or any inactive excipient of the study drug.
* Women who are breastfeeding.
* With alcohol or drug abuse disorder.
* History of stroke or intracranial hemorrhage with 6 months prior to screening.
* Attenuated live vaccination within 4 weeks prior to screening.
* With basic medical condition leading to risk of taking study drugs judged by investigators, or with confusion to toxicity and adverse events.
* Judgment by the investigator that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2020-05-09 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 12 months
  Proportion of patients who have either a complete or partial response before any treatment change.
Lymph Node Response (LNR) | up to 12 months
  LNR was defined as the percentage of participants who achieved a ≥ 50% decrease from baseline in the sum of the product of the perpendicular diameters (SPD) of measurable index lesions.
Time to Response (TTR) | up to 12 months
  TTR was defined as the interval from the start of SHC014748M treatment to the first documentation of complete response(CR) or partial response(PR).
Progression-Free Survival (PFS) | up to 12 months
  PFS was defined as the interval from the start of SHC014748M treatment to the earlier of the first documentation of disease progression or death from any cause. PFS was analyzed using Kaplan-Meier (KM) estimates.
Duration of Response (DOR) | up to 12 months
  DOR was defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of disease progression as or death from any cause. DOR was analyzed using KM estimates.
Mean Change From Baseline in the Functional Assessment of Cancer Therapy Lymphoma (FACT-Lym) Scale. | up to 12 months
  The FACT-Lym questionnaire is a validated instrument for assessing the impact of lymphoma on health related quality of life(HRQL) and contains 42 questions covering HRQL and common lymphoma symptoms and treatment side-effects. It begins with the Functional Assessment of Cancer Therapy - General (FACT-G), which contains 27 questions covering four core subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The FACT-Lym also includes an Additional Concerns subscale (15 questions) used to assess non-Hodgkins lymphoma(NHL) related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). Higher scores are associated with a better quality of life.

SECONDARY OUTCOMES:
Safety and Tolerability of SHC014748M Assessed as the Number of Participants Experiencing Adverse Events (AEs) or Abnormalities in Vital Signs, Laboratory Tests, or Electrocardiograms. | up to 12 months
Pharmacokinetics Parameter: Cmax | 4 weeks
Pharmacokinetics Parameter: Tmax | 4 weeks
Pharmacokinetics Parameter: ACUlast | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No